CLINICAL TRIAL: NCT03752697
Title: Longitudinal Examination of Metacognition in Neurological Samples
Brief Title: Metacognition in Neurological Injury
Status: Active, not recruiting | Type: Observational
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Quality Living, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18123
Record Dates: First submitted 2018-09-25; First posted 2018-11-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Brain Injuries
Keywords: metacognition; self-assessment
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurological injury: Paper and pencil/computerized assessments of cognitive functioning and metacognitive performance will be administered.
  Interventions: Behavioral: metacognitive performance
- Healthy control: Paper and pencil/computerized assessments of cognitive functioning and metacognitive performance will be administered.
  Interventions: Behavioral: metacognitive performance

INTERVENTIONS:
Behavioral: metacognitive performance — Paper and pencil/computerized tests of metacognition

SUMMARY:
The purpose of this study is to investigate the trajectory of metacognitive functioning throughout phases of recovery from neurological insult, and to determine its relationship to rehabilitation compliance and functional outcome. It is hypothesized that metacognitive accuracy improves over time, and is a significant predictor of engagement in rehabilitation activities.

DETAILED DESCRIPTION:
This study will examine the trajectory of metacognitive functioning through different phases of recovery from neurological insult, and document its relationship to rehabilitation compliance. Individuals currently completing rehabilitation programs and individuals from the community who meet study criteria are invited to participate. After consenting and enrolling in the study, participants complete 2 study sessions: a baseline session, and a follow-up session either at time of completion of rehabilitation program or 3 months later if not in a rehabilitation program. During the study sessions, participants will complete paper-and-pencil and computerized tests of cognition (including metacognitive tasks).

ELIGIBILITY:
Inclusion Criteria:

* history of brain and/or spinal cord injury
* no history of brain or neurological injury/insult (for healthy control group)
* fluent in spoken and written English
* adequate gross motor abilities to provide a button push on a keyboard

Exclusion Criteria:

* exclusion criteria for healthy controls include:
* current/past history of psychiatric illness
* learning disorder
* developmental disorder
* diagnosis of Attention Deficit Disorder/Attention Deficit Hyperactive Disorder

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants in rehabilitation facility and community-dwelling individuals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline metamemory performance to completion of rehabilitation | At baseline and at end of length of stay in rehabilitative setting (on average 3 months)
  The computerized metamemory test produces scores that are used to calculate a gamma coefficient, which is a quantitative measure of the individual's metacognitive performance/accuracy.

SECONDARY OUTCOMES:
Change in rehabilitative engagement | At baseline and at end of length of stay in rehabilitative setting (on average 3 months)
  The rehabilitative engagement questionnaire is a clinician-report measure that queries the clinician's perception of their client's participation in rehabilitation services.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Chiou, Ph.D., Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No